CLINICAL TRIAL: NCT03320343
Title: Pilot Study of Measurement Agreement Between Morphological and Diffusion Tensor Imaging MRI for Pelvic Nerve Cartography
Acronym: NERVWATCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2017-01/MB-01
Record Dates: First submitted 2017-10-17; First posted 2017-10-25 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Pelvic MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients recruited for pelvic imaging examination
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — 3D morphological MRI and diffusion tensor imaging

SUMMARY:
The investigators hypothesize that diffusion tensor imaging (DTI) will produce a similar map of autonomic pelvic innervation to that obtained using 3D morphological MRI sequences

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient it at least 18 years old
* The patient has been admitted for an MRI examination of the pelvic region, for any reason

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant or breast feeding
* There is a contra-indication for MRI (pacemaker, claustrophobic patient)
* The patient has had previous pelvic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Medical Imaging Department of the CHU Nîmes for an MRI examination of the pelvic region for any reason
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Agreement between DTI imaging measures versus 3D morphological MRI measures for point of penetration of the pelvic splanchnic nerves in the lower hypogastric plexus | Day 0
  Lin's concordance correlation coefficient and Bland-Altman Plot
Agreement between DTI imaging measures versus 3D morphological MRI measures for point of penetration of the pelvic hypogastric nerves in the lower hypogastric plexus | Day 0
  Lin's concordance correlation coefficient and Bland-Altman Plot
Agreement between DTI imaging measures versus 3D morphological MRI measures for origin of the cavernous nerves | Day 0
  Lin's concordance correlation coefficient and Bland-Altman Plot

SECONDARY OUTCOMES:
Acquisition time | Day 0
  min
Time necessary for sequence reconstruction | Day 0
  min
Inter-operator agreement | Day 0
  Kappa coefficient of measurements between two operators
Intra-operator agreement | Month 6
  Kappa coefficient of measurements from same operator 6 months apart

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nimes, Nîmes, France